CLINICAL TRIAL: NCT01318681
Title: Effects of Treated and Untreated Allergic Rhinitis on Mood, Cognitive Functions and Actual Driving Performance
Brief Title: Rhinitis, Cognition and Driving Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Vuurman, DR Eric Vuurman, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: EPU-055; NCT01239264 (obsolete NCT alias)
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2011-03

CONDITIONS: Seasonal Allergic Rhinitis; Driving Ability; Cognition
Keywords: driving, memory, cognition
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Cetirizine; fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pollen provocation with systemic treatment (Experimental): Subjects are treated with Cetirizine 10 mg after a nasal challenge with a pollen solution
  Interventions: Drug: cetirizine 10 mg
- Pollen provocation with topical treatment (Experimental): treatment with 25ug fluticasone furoate after a nasal pollen challenge
  Interventions: Drug: fluticasone furoate
- placebo treatment after pollen challenge (Placebo Comparator): Placebo treatment after a nasal challenge with pollen solution
  Interventions: Drug: placebo
- control condition (No Intervention): A placebo drug is administered after a sham nasal challenge with a pollen solution

INTERVENTIONS:
Drug: cetirizine 10 mg — cetirizine 10 mg over encapsulated
  Arms: Pollen provocation with systemic treatment
Drug: fluticasone furoate — nasal spray 25ug per dose
  Arms: Pollen provocation with topical treatment
Drug: placebo — a placebo nasal spray and placebo capsule are available for double dummy treatment
  Arms: placebo treatment after pollen challenge

SUMMARY:
This study investigates the effects of Allergic Rhinitis (AR) on driving ability and memory functions. Our group has previously shown that patients suffering from AR symptoms perform less well on tasks requiring sustained attention compared to non symptomatic controls. Car driving is a typical behavior that is susceptible for changes in sustained attention and might therefore become worse under conditions when patients suffer from AR symptoms. We will compare the driving performance of untreated, symptomatic AR patients with the performance of symptomatic patients that have been treated with either a systemic AR medication (a pill) or a topical medication (nasal spray)

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers known with Seasonal Allergic Rhinitis
* Experienced drivers holding a license
* 21- 45 years of age

Exclusion Criteria:

* Asthma or other chronic illness
* current psychoactive medication
* History of drug abuse

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP) in highway driving | 2:00 - 3:00 hrs post dosing
  Standard Deviation of Lateral Position (SDLP) is the amount of "weaving" that occurs when a person is driving in a straight line on the highway and instructed to maintain a steady speed and position within the lane he/she is driving

SECONDARY OUTCOMES:
Word Learning Test (WLT-15) verbal memory score | 2:30 hrs post dosing
  Subjects are presented with a list of 15 words at a rate of one word/second with a pause between words of one second. Immediately following the presentation subjects are asked to recall and name as many words as possible. The total number of words recalled after three repeated presentations of the same list of words is the outcome variable

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands